CLINICAL TRIAL: NCT00333710
Title: Evaluating a Telehealth Treatment for Veterans With Hepatitis C and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: F4120-V
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Disease; Hepatitis C; Stress Disorders, Post-Traumatic
Keywords: Rehabilitation; Telecommunication
MeSH Terms: conditions — Chronic Disease; Hepatitis C; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual face-to-face contact (Experimental): Individual face-to-face contact treatment
  Interventions: Behavioral: Individual psychotherapy
- Individual telephone contact (Experimental): Individual telephone contact treatment
  Interventions: Behavioral: Telehealth Intervention
- Control condition/treatment as usual (No Intervention): Control condition/treatment as usual

INTERVENTIONS:
Behavioral: Individual psychotherapy — Individual face-to-face contact with educational and goal setting components
  Arms: Individual face-to-face contact
Behavioral: Telehealth Intervention — Individual telephone contact with educational and goal setting components
  Arms: Individual telephone contact

SUMMARY:
The main objective of this proposal is to develop and test the efficacy of two interventions (a telehealth and face-to-face intervention) designed to improve quality of life, self-care, motivation to engage in healthcare, and psychological distress in patients diagnosed with HCV and PTSD. It is hypothesized that

DETAILED DESCRIPTION:
Patients with comorbid diagnoses of HCV and PTSD may experience increased risk of diminished quality of life, given that PTSD is associated with poor self-care and medical non-compliance. To date, no systematic efforts to improve quality of life in this high-risk population have been documented. The main objective of this proposal is to develop and test the feasibility and efficacy of two cognitive-behavioral interventions (a telehealth intervention and a face-to-face intervention) designed to improve quality of life, self-care, motivation to engage in healthcare, and psychological distress in patients diagnosed with HCV and PTSD. A secondary objective is to evaluate the cost effectiveness of the interventions. I plan to develop the interventions, pilot test them, and deliver the refined treatments to veterans with HCV and PTSD. Participants will be 70 patients from VA Boston who meet study criteria. Assessment will occur at pre-treatment, post-treatment, and 3- and 6-month follow-up. Assessments will measure quality of life, self-care, motivation to engage in healthcare, and psychological distress. Analyses will examine study feasibility, the effects of the treatment conditions, and the cost effectiveness of the interventions. It is hypothesized that the telephone and face-to-face intervention will improve outcomes, as compared to treatment as usual, but that the participants will be more satisfied with the telephone intervention. In addition, it is predicted that the telephone condition will be cost effective as compared to the face-to-face intervention

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatitis C
* Clinical diagnosis of posttraumatic stress disorder
* Need to have access to a telephone

Exclusion Criteria:

* Life threatening or acute illness
* Current alcohol or substance dependence
* Currently prescribed interferon treatment
* No access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Silberbogen, PhD, Principal Investigator — VA Medical Center, Jamaica Plain Campus
Locations (1):
- VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individual Face-to-face Contact | Individual Telephone Contact | Control Condition/Treatment as Usual
Started | 19 | 18 | 16
Completed | 8 | 14 | 15
Not Completed | 11 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Condition/Treatment as Usual: Control condition/treatment as usual.
  No active treatment
- Total: Total of all reporting groups
Arm/Group | Individual Face-to-face Contact | Individual Telephone Contact | Control Condition/Treatment as Usual | Total
Number analyzed (Participants) | 19 | 18 | 16 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.37 (4.89) | 52.28 (5.19) | 55 (6.80) | 53.85 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4
  Male | 16 | 17 | 16 | 49
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 16 | 53

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis C Virus Knowledge Questionnaire
Description: This is a 62-item measure which assesses knowledge of the hepatitis C Virus. Range is 0 to 62. Higher scores reflect greater hepatitis C knowledge
Time Frame: pre-treatment, post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Face-to-face Contact | Individual Telephone Contact | Control Condition/Treatment as Usual
Number analyzed (Participants) | 8 | 14 | 15
units on a scale
  Pre-Treatment | 37.88 (10.78) | 40.50 (6.19) | 35.80 (10.05)
  Post-Treatment | 45.38 (7.89) | 42.36 (6.03) | 34.73 (11.09)

ADVERSE EVENTS:
Time Frame: During recruitment and when running subjects
Arm/Group | Individual Face-to-face Contact | Individual Telephone Contact | Control Condition/Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
Small sample size, all male, reliance on self-report measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes